CLINICAL TRIAL: NCT07397000
Title: Development of AI-Based Approaches for Automated Real-Time Detection of Surgical Smoke Using Endoscopic Image and Video Data
Brief Title: AI-Based Real-Time Detection of Surgical Smoke Using Endoscopic Data
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: MT_STORZ Rauchgasabsaugung
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Detection of Surgical Smoke Gas Using AI

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational, prospective monocentric pilot study is to generate a pilot dataset to train a computer-assisted model for automatic, intraoperative detection of surgical smoke gas.

Women with indications for laparoscopic evaluation requiring the use of HF surgery (expecting the formation of smoke gas) and a smoke evacuation system (Karl Storz S-Pilot) are employed.

DETAILED DESCRIPTION:
Detection of surgical smoke gas with an accuracy F1 score of >= 0.8 on test datasets. The activation of the S-Pilot by clinic personnel will be used as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 years
* Written consent after receiving information
* Indication for surgical treatment using HF surgery

Exclusion Criteria:

* - Expected lack of compliance by the patient or inability of the patient to understand the meaning and purpose of the clinical trial
* Lack of patient consent
* S-Pilot cannot be used

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years or older undergoing laparoscopic gynecological procedures at the Department of Women's Health, University Hospital Tübingen, where high-frequency surgical technology (monopolar, bipolar, or ultrasound) is used and surgical smoke generation is expected. All procedures will utilize the KARL STORZ S-Pilot smoke evacuation system.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Detection of surgical smoke gas | At the end of the study (9 months)
  Detection of surgical smoke gas with an accuracy of an F1 score of ≥ 0.8 on test data sets.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Bernhard Krämer, Principal Investigator — Deparment of Women's Health, University Hospital Tübingen
Locations (1):
- Department of Women's Health, University Hospital, Tübingen, Germany